CLINICAL TRIAL: NCT01640899
Title: The Effect of Shoe Insoles on Pain and Daily Activities and the Relation Between Satisfaction With Insoles and Use: A pre-and Post-intervention Survey
Brief Title: Insoles Effect on Pain and Daily Activities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Rehabilitation Research, Örebro (Other Government)
Collaborators: Örebro County Council (Other Government)
Responsible Party: Principal Investigator, Ahmed Amer, Research Assisstant, Centre for Rehabilitation Research, Örebro
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRR120709
Record Dates: First submitted 2012-07-12; First posted 2012-07-16 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Non-specific Pain in Lower Extremities
Keywords: Orthotic Devices; Activities of Daily Living; Pain Measurement; Lower Extremity; Foot; Personal Satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single-arm study (Other): This is a single-arm study. Just one group (i.e. the patients)
  Interventions: Device: Shoe Insoles

INTERVENTIONS:
Device: Shoe Insoles — Shoe insoles is an orthotic devices which are used to prevent, relieve, or reduce pain in lower extremities. The insoles give a mechanical support for the body by put it in a good alignment.

SUMMARY:
The aims of this study were to evaluate the effects of insoles on pain, daily activities and physical activity level, and to investigate the relation between satisfaction with the insoles and their actual use in individuals with LE pain.

DETAILED DESCRIPTION:
Pain in weight-bearing joints limits individual's function and ability to perform daily activities, causes a negative effect on productivity and increased costs for social insurance. This pain is often the outcome of structural deformities or work-related foot pain often occurs in workers whose occupations include standing or walking for a long time.

One of the most common reasons for prescribing insoles is to enhance functioning by reducing nonspecific pain in the foot, leg or low back pain. Reduction of pain is expected to improve quality of life in daily activities such as work and recreational activities.

Persons actual use of the insoles, is a prerequisite for any effect it may have. It can be hypothesized that the use of the insoles is related to what the user thinks about their comfort, appearance, the amount of foot perspiration they induce, and other factors.

ELIGIBILITY:
Inclusion Criteria:

* Pain in lower extremities
* Aged 18 years or older
* Able to speak Swedish.

Exclusion Criteria:

* Pain due to a systemic or progressive disease
* Use of orthosis of other type than insoles
* Earlier foot surgery or current use of prosthesis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2010-08; Primary Completion 2011-01 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Shoe insoles effect on pain level in lower extremities. | Four-weeks follwo up period
  The participants answer the inetial questioniners before getting the insoles, then answr the same questionnier after four weeks of insoles use.
Shoe insoles effect on daily activities | Four-weeks follow up period
  The participants answer Inetnational Physical Activty Questionnier (IPAQ)and Lower Extremity Functional Status (LEFS)before getting the insoles and after four weeks of use.
Satisfaction with shoe insoles use | After four weeks of use
  Client Satisfaction with Device(CSD)survey was anwered by the participants after four weeks of use.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Amer, Master, Principal Investigator — Centre for Rehabilitation Reserach, Örebro; Liselotte Norling-Hermansson, PhD, Study Director — Dept. of Prosthetics and Orthotics, Örebro University Hospital, Örebro
Locations (1):
- Dept. of Prosthetics and Orthotics, Orebro University Hospital, Örebro, Örebro County, Sweden

REFERENCES:
- See also: Information about the study (In Swedish) — http://www.orebroll.se/sv/Forskning/Forskningsomraden/HFC1/personalHFC/Ahmed-Amer/Examensarbete-Ahmed-Amer/
- See also: Main page of Centre for Rehabilitation Research — http://www.orebroll.se/en/Research/Forskningsomraden/Information-in-English/